CLINICAL TRIAL: NCT02130102
Title: Evaluation of ModuLAAr - a Module Based and Scalable System for Silver-ager Located in Assisted Living Homes in Austria
Brief Title: ModuLAAr - A Module Based and Scalable System for Silver-ager in Austria
Acronym: ModuLAAr
Status: Completed | Type: Observational
Sponsor: AIT Austrian Institute of Technology GmbH (Other)
Collaborators: Samariterbund Burgenland Rettung und Soziale Dienste GmbH (Unknown); University of Applied Sciences Technikum Wien (Unknown); Austrian Research Promotion Agency (Other Government); Austrian Federal Ministry of Transport, Innovation and Technology (BMVIT) (Unknown)
Responsible Party: Principal Investigator, Christian Siegel, Research Associate, AIT Austrian Institute of Technology GmbH
Other Study IDs: FFG Registration Nr. 835863
Record Dates: First submitted 2014-04-30; First posted 2014-05-05 (Estimated); Last update posted 2015-12-31 (Estimated); Status verified 2015-12

CONDITIONS: Quality of Life
Keywords: technology acceptance; ambient assisted living; independent living; quality of life; socioeconomic impact; usability of information and communication technologies

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Users of ModuLAAr: A group of volunteers (aged 60+), living in assisted living homes, will be provided with module based technical solutions to improve their independency and quality of life.
  Interventions: Device: The ModuLAAr Ambient Assisted Living System

INTERVENTIONS:
Device: The ModuLAAr Ambient Assisted Living System — The system consists of the following modules which will be provided to the volunteers according to their needs:
  tablet computer (digital photo album, video telephone, meal ordering system, reminder system), bodyweight scale, blood pressure meter, emergency call system, mobile phone (documentation of personal health-related data), bathroom surveillance system, blood glucose meter, house automation technologies/smart home technologies

SUMMARY:
In this research project a module based Ambient Assisted Living solution will be provided to elderly living in assisted living homes. Those products and services seek to impact quality of life of the elderly and have positive effects on their environment.

ELIGIBILITY:
Inclusion Criteria:

* 60 years and older
* informed consent
* resident of an assisted living home of the Samariterbund Burgenland Rettung und Soziale Dienste GmbH

Exclusion Criteria:

* relevant health threatening event or death
* mini mental state score <17

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: elderly residents of assisted living homes aged 60 and above
Sampling Method: Non-Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2013-06; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Changes of quality of life and subjective health | 4 and 1 months before intervention. 1, 4 and 12 months after intervention
  multidimensional outcome assessment of quality of life: Quality of life is assessed by the questionnaires of the World Health Organization (WHOQOL-BREF and WHOQOL-OLD) as well as with semi-structured qualitative interviews. Subjective health is assessed by EQ-5D VAS of the Euroqol-Organization.

SECONDARY OUTCOMES:
Changes in technology acceptance and usability | 1, 12 and 18 months after intervention
  qualitative evaluation according to the technology acceptance model (TAM) and usability questionnaire
Impact and changes on socio-economic parameters | 4 months before intervention. 4 and 12 months after intervention
  user-questionnaire with socio-economic and socio-demographic parameters: (gender, income, housing conditions, level of education, level of social support, working experience, medicine intake, chronic diseases, frequency of falls, health threatening events).
  Semi-structured qualitative interviews using the delphi method will be conducted.

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Prazak-Aram, Mag., Principal Investigator — AIT Austrian Institute of Technology GmbH
Locations (1):
- AIT Austrian Institute of Technology GmbH, Wiener Neustadt, Lower Austria, Austria

REFERENCES:
- [Derived] Siegel C, Prazak-Aram B, Kropf J, Kundi M, Dorner T. Evaluation of a modular scalable system for silver-ager located in assisted living homes in Austria--study protocol of the ModuLAAr ambient assisted living project. BMC Public Health. 2014 Jul 21;14:736. doi: 10.1186/1471-2458-14-736. PMID 25047720
- See also: Website of the ModuLAAr project — http://www.modulaar.at